CLINICAL TRIAL: NCT01625975
Title: A Retrospective Study to Assess the Outcome After Treatment With the Eight Plate System in Pediatric Patients
Brief Title: Retrospective Eight Plate Study
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: 106309
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Leg Length Discrepancy; Varus/Valgus Deformities of the Knee
Keywords: Growth modulation; Eight plate; Leg length discrepancy; Varus/valgus deformities; Pediatric
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Growth modulation with Eight plate: Pediatric patients undergoing growth modulation with the Eight plate system

SUMMARY:
Understanding bone growth and achieving bone deformity corrections re-mains one of the oldest challenges in paediatric orthopaedics.

The purpose of this study is to investigate the clinical and biomechanical effects of implants for growth modulation in pediatric patients undergoing correction of leg length or deformities of the knee.

The primary aim of the study is to assess outcome after growth modulation using the Eight plate (Orthofix) at the time of implant removal with regard to any Adverse Events (AE) related to the growth plates or implants under investigation. The secondary aims are to assess if the planned correction was achieved and if the achieved correction was maintained after implant removal. Furthermore, secondary aims include investigation of the number and type of revision surgeries, the proportions of any other local AE as well as any influencing factors for growth modulation.

DETAILED DESCRIPTION:
One of the oldest mysteries in paediatric orthopaedics is the knowledge about bone growth and the ability to correct acquired bone deformities. Guiding the growth of a bone for deformity cor-rection by harnessing the ability of a growing bone to undergo plastic deformity is a well-known pediatric orthopaedic principle. Nevertheless, there are still many open questions concerning growth and guided growth. Several surgical options already exist for correction of angular de-formity and leg length discrepancies. The gold standard remains the corrective osteo¬tomy before or after growth arrest.

Correction during growth poses the risk of recurrence of the deformity during growth. By any means, growth modulation involves major surgery and requires internal or external fixation. Epiphysiodesis or hemiepiphysiodesis, either permanent or temporarily, can be done in an open or percutaneous way. Permanent epiphysiodesis is mainly performed using screws, while for a temporary epiphysiodesis staples or plate/screw systems are used. The treatment seems to be clinically effective, but the precise calculation of the remaining growth and the optimal surgical timing are crucial. Furthermore, the underlying biomechanical properties are not yet fully known.

The objective of this study is to investigate the clinical effects of the Eight Plate system for growth modulation treatments in pediatric patients undergoing leg length corrections or deformity corrections of the knee. The primary aim of the study is to assess outcome of growth modulation at removal of the implants with regards to AEs related to the growth plates or implants under investigation. The secondary aims are to assess if the planned correction was achieved and if the achieved correction was maintained after Eight Plate removal. Furthermore, secondary aims include the investigation of the number and type of revision surgeries, any functional deficits after implant removal, any additional local AE, the assessment of the primary implant positioning, and any additional radiological parameters related to the implants and leg alignment.

ELIGIBILITY:
Inclusion Criteria:

* Age range at implantation of the Eight Plate growth modulation devic-es: 18 months to 17 years
* Treatment with Eight Plate (Orthofix) of varus/valgus deformities of the knee and/or leg length discrepancy due to any of the following:
* Diseases or syndromes affecting the growth plate (eg, Blount's dis-ease)
* Post-traumatic, affecting the growth plate
* Post-infectious, affecting the growth plate
* Idiopathic etiology
* Documented implantation of Eight Plate system(s) within the last 5 years
* Documented explantation of all Eight Plate system(s)
* Able to walk without walking aids prior to Eight Plate implantation

Exclusion Criteria:

* Any tumor possibly influencing the growth plate(s) prior to last follow-up visit considered for this study
* Cerebral palsy

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with an age range at implantation of the Eight Plate growth modulation devices of 18 months to 17 years
  Treatment with Eight Plate (Orthofix) of varus/valgus deformities of the knee and/or leg length discrepancy due to any of the following:
  * Diseases or syndromes affecting the growth plate (eg, Blount's dis-ease)
  * Post-traumatic, affecting the growth plate
  * Post-infectious, affecting the growth plate
  * Idiopathic etiology
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theddy Slongo, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (7):
- Germany (2):
  - Kinderchirurgische Klinik Städtisches Klinikum Karlsruhe, Karlsruhe
  - Klinikum Stuttgart, Stuttgart
- Sancheti Institute for Orthopaedics and Rehabilitation, Pune, India
- Switzerland (3):
  - Inselspital Bern, Bern
  - Hôpital des enfants, Geneva
  - Universitätskinderspital Zürich, Zurich
- Guy Hilton Research Centre ISTM, Keele University, Stoke-on-Trent, United Kingdom